CLINICAL TRIAL: NCT07159633
Title: OurRelationship-S: A Digital Relationship-Strengthening Program for Couples Experiencing Substance Misuse
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OurRelationship (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SUD SBIR Phase 1; R43DA059979-01A1 (NIH)
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Relationship Conflict; Relationship Distress
Keywords: OurRelationship; Couples; Digital; Online; Recovery; Substance use disorder
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Couples in the Experimental arm receive the 8-hour online OurRelationship program plus six 20-minute calls with a project coach.
  Interventions: Behavioral: Online Couple Intervention

INTERVENTIONS:
Behavioral: Online Couple Intervention — The OurRelationship program is approximately 8-10 hours of online content and will delivered over the course of 5-8 weeks. For the current study, we have tailored the general OurRelationship content for couples in recovery from substance misuse. For example, all users receive informational material on the nature of addition and recovery. All of the videos in the adapted program depict couples struggling with recovery-related issues. Additionally, the assessments and feedback content has been tailored. In addition to the online content, couples receive up to 100 minutes of scheduled coach Zoom calls (up to five 20-minute calls).
  Other Names: OurRelationship; Our Relationship

SUMMARY:
This study tests the effectiveness of an online relationship program that has been tailored for couples in which one or both members are in recovery from substance misuse. The purpose of this program is to strengthen the romantic relationship and improve individual functioning. Couples participate in approximately 8 hours of digital content (on their phone or computer) and have a total of five calls with a project coach. Couples will be asked to complete online surveys before and after the program and are paid $200 per couple ($100 per individual) for doing so.

DETAILED DESCRIPTION:
Relationship conflict and distress are common presenting complaints during recovery from SUD and can lead to a reoccurrence and/or increase in use of substances. Poor romantic relationships also interfere with successful SUD treatment and recovery interventions. Therefore, documenting the effects of the initial version of the Our Relationship program tailored for couples in recovery and generating ideas for subsequent improvements will be important advancements in efforts to increase social recovery capital for individuals with substance misuse.

The OurRelationship program is based on the empirically-supported Integrative Behavioral Couple Therapy (IBCT) approach, which has been found to have beneficial effects through five years after treatment. IBCT was translated into a web-based format by Dr. Brian Doss. As part of a completed R01-funded project, 300 couples were randomly assigned to receive the OurRelationship program or to a wait-list control group (Doss et al., 2016). Compared to the waitlist group, intervention couples reported significant improvements in relationship satisfaction (Cohen's d = 0.69), relationship confidence (d = 0.47), and negative relationship quality (d = 0.57). Additionally, couples reported significant improvements in multiple domains of individual functioning, especially when individuals began the program with difficulties in that domain: depressive (d = 0.71) and anxious symptoms (d = 0.94), perceived health (d = 0.51), work functioning (d = 0.57), and quality of life (d = 0.44).

In another completed RCT (Doss et al., 2020; Roddy et al., 2020), almost 2,000 low-income couples were randomly assigned to receive the Our Relationship program or a wait-list control group. Compared to the waitlist control group, those that received the OurRelationship program experienced improvements in relationship satisfaction (d = 0.53), emotional support (d = 0.46), as well as decreases in breakup potential (d = -0.53), conflict (d = -0.78), and the presence of IPV (d = -0.10). Most notably for the present study, participants who reported problematic alcohol use at baseline experienced significantly greater reductions in problematic alcohol use than did those in the control group (d = -0.33).

Recruitment

Couples will be recruited from five community recovery organizations that have agreed to partner in this project. As part of their standard intake process, Our-S will be offered to all appropriate individuals (e.g., those in a committed romantic relationship of at least 6 months duration). Clients will be provided with pamphlets to deliver to their partner as well as a dedicated webpage designed to address partner-perspective questions and concerns.

Description of the OurRelationship program:

The OurRelationship program is approximately 8-10 hours of online content and will delivered over the course of 5-8 weeks. In this program, partners complete the majority of the program on their own (to make it more flexible) and come together for 2-3 key conversations with their partner. The first section of the program, "Observe", helps individuals in brainstorming potential relationship problems on which to focus. The first conversation between partners centers on discussing possible core relationship issues and jointly deciding on the problem(s) to focus on during the program. The "Understand" section leads the individual through steps to achieve a more accurate understanding of the problem, including how differences between partners, hidden emotions, external stressors, and patterns of communication might affect the core issue(s). During the two "Understand" conversations, both partners' previous written responses are displayed on the screen and conversation is encouraged. The "Respond" phase, to help partners develop a plan for fixing the problem, includes information about acceptance and self-change, communication tips, and suggestions tailored to their presenting problem. During the "Respond" conversation, couples share their strategies to decrease stress, improve patterns of communication, and engage in problem-solving exercises specific to their core issue(s). Throughout the program, screens include combinations of text, audio, still graphics, and videos. Four example couples, representing African-American, Hispanic, and White couples, are followed through the program. Other screens present interactive graphs based on how users answered questions, such as showing whether they report higher or lower stress than average. Users also receive tailored text feedback on their scores.

For the current study, the general OurRelationship content was tailored for couples in recovery from substance misuse. For example, all users will view informational material on the nature of addition and recovery. All of the videos in the adapted program depict couples struggling with recovery-related issues. Additionally, the assessments and feedback content has been tailored. For example, in the Differences chapter, couples see how they and their partner score on sensation seeking as well as anxious and avoidant attachment. Similarly, in the Stress chapter, users view common stressors (misuse-linked money problems, lingering physical and mental health effects) related to recovery from substance misuse.

In addition to the online content, couples will receive up to 100 minutes of scheduled coach calls (up to five 20-minute calls). These coach calls will either occur via Zoom a phone call - as selected by the couple. These calls occur before the program, during the program, and at the end of the program.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate, couples will need to be:

1. in a romantic relationship and married, engaged, cohabiting, or dating exclusively for >6mo;
2. Age 18+
3. Both partners are willing to participate in the study
4. Both partners are fluent readers of the English language and
5. One or both members of the couple are currently in treatment or recovery services for substance use-related issues.

Exclusion Criteria:

1. Severe domestic violence: We will utilize exclusion criteria for domestic violence that we have used for the last seven years of OurRelationship services with low-income and military couples. These criteria were developed in consultation with CEO of the National Resource Center on Domestic Violence and several members of the Domestic Violence Hotline. Through these conversations, we concluded it would be appropriate if couples were excluded from OurRelationship services if either person reports in the past 6 months that their partner: 1) Choked me 2) Repeatedly punched me during a fight or beat me up 3) Threatened me with (or used) a gun or knife, or 4) Physically forced me to have sex when I didn't want to. Finally, couples will be excluded if either person reports in the past 6 months that: 5) he/she was "quite afraid", "very afraid", or "extremely afraid" that their partners would physically hurt them during an argument.
2. Inadequate internet connection. To ensure that the program can function properly, participants will be required to have access to high-speed internet in their homes or on their smartphones (with regular wireless/hotspot or a minimum 4G cellular connection).
3. Have already decided to end the relationship. Because the tested programs are designed to help couples improve their relationships (rather than deal with a separation or divorce), couples will be excluded if either partner endorses that they "will probably end my relationship even if it does get better" or that they "have already made the decision to end my relationship."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship satisfaction | From enrollment to the end of the program (or point of dropout) - approximately 8 weeks later.
  Global relationship satisfaction, measured by the 8-item version of the Couple Satisfaction Index (CSI-8) will be used to assess changes during the program. Scores range from 0-41, with higher scores indicating more satisfaction
Relationship conflict | From enrollment to the end of the program (or point of dropout) - approximately 8 weeks later.
  This 5-item measure captures the frequency of arguments, criticism, and disrespectful behavior in the previous month on a Likert scale. Scores range from 5-20, with higher scores indicating more conflict.

SECONDARY OUTCOMES:
Emotional trust | From enrollment to the end of the program (or point of dropout) - approximately 8 weeks later.
  This 5-item, Likert-scale subscale has been shown in our studies to mediate subsequent improvements in relationship satisfaction. Scores range from 5-20, with higher scores indicating more trust.
Relational recovery capital | From enrollment to the end of the program (or point of dropout) - approximately 8 weeks later.
  The 10-item Social Support subscale of the Assessment of Recovery Capital (ARC) will be used to determine whether effects generalize to friends and family. Scores range from 10-60, with higher scores indicating more social support.
Program Evaluation | From enrollment to the end of the program (or point of dropout) - approximately 8 weeks later.
  The 8-item Client Evaluation of Services Questionnaire has been administered in previous studies of OurRelationship and BCT, providing a useful comparison. Scores range from 8-32, with higher scores indicating greater satisfaction with services.

CONTACTS AND LOCATIONS:
Overall Officials: Brock Sansbury, MBA, Principal Investigator — OurRelationship LLC; Brian D Doss, Ph.D., Study Director — OurRelationship LLC
Locations (5):
- United States (5):
  - Innovia Behavioral Health, Marietta, Georgia
  - Voices of Hope Maryland, Elkton, Maryland
  - Commonly Well, Potsdam, New York
  - The Courage Center, Lexington, South Carolina
  - Youturn Health, Coppell, Texas

IPD SHARING:
Plan to Share IPD: Yes
We will provide a de-identified dataset consisting of key demographics, primary and secondary outcome measures, and information on program completion.
Supporting Information: Study Protocol, ICF
Time Frame: The IPD file will be available 6 months after the end of the trial and will be available for at least two years.
Access Criteria: Data will be available to qualified researchers. Please email the PI, Brock Sansbury, at brock@ourrelationship.com

REFERENCES:
- See also: Enrollment site for participants — https://www.ourrelationship.com/recovery